CLINICAL TRIAL: NCT03789227
Title: CT-guided Ethyl Alcohol Ablation of the Ganglion Impar for Pelvic Tumors: Does the Addition of Ketorolac or Dexamethasone Makes a Difference?
Brief Title: CT-guided Ablation of the Ganglion Impar for Pelvic Tumors: Comparethe Addition of Ketorolac or Dexamethasone
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mansoura University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: - MFM-IRB ,MD ∕ 16.06.45
Record Dates: First submitted 2018-12-26; First posted 2018-12-28 (Actual); Last update posted 2020-09-03 (Actual); Status verified 2020-09

CONDITIONS: Pain, Chronic
MeSH Terms: conditions — Chronic Pain

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Group C (Placebo Comparator): ganglion impar block :patients will receive a premixed solution of 3 ml lidocaine 2%, 5 ml absolute alcohol 95% and 4 ml saline in a total volume 12 ml.
  Interventions: Procedure: ganglion impar block
- Group D (Active Comparator): ganglion impar block :patients will receive a premixed solution of 3 ml lidocaine 2%, 5 ml absolute alcohol 95% and 8 mg dexamethasone with 4 ml saline in a total volume 12 ml.
  Interventions: Procedure: ganglion impar block
- Group K (Active Comparator): ganglion impar block :patients will receive a premixed solution of 3 ml lidocaine 2%, 5 ml absolute alcohol 95% and 15 mg ketorolac with 4 ml saline in total volume 12 ml.
  Interventions: Procedure: ganglion impar block

INTERVENTIONS:
Procedure: ganglion impar block — the patient will be in the prone position with a pillow under the abdomen The pre-injection planning images will be obtained using CT with 2 mm axial section thickness. Under aseptic technique, a skin wheal will be raised with 2 ml lignocaine 0.5% using 23 G needle either in midline or paramedian approach. After identifying the ganglion impar, usually at the level of the sacro-coccygeal disc, a 25 G, 9 cm long spinal needle will be introduced at approximately 6-9 cm from midline and a small amount of non-ionic contrast medium (0.5 ml iopamidol; 300 mg/ml) will be injected. The midline approach may be selected according to patient position and operative condition. In the midline approach the sacro-coccygeal disc is identified and needle will be introduced perpendicular through the disc and just encroaching upon presacro-coccygeal space. Thereafter, 3 ml lidocaine 2% will be injected, three minutes later 5 ml absolute alcohol 95%.

SUMMARY:
this study investigator will resaearsh about the efficacy of addition of ketorlac or dexamethasone to alcohol in ablation of ganglion impar in pelvic tumour to asses thier efficacy in increasing the intensity or the duration of the block

DETAILED DESCRIPTION:
The aim of this study is to compare the effect of administration of ketorolac versus dexamethasone on CT guided ganglion impar block with ethyl alcohol in patients with pelvic tumor.

The primary outcome will be the onset of sensory block, patient satisfaction measured by patient satisfaction score ( Jones KD, Sutton C., 2003), intensity of pain measured by a linear visual analogue scale (VAS) (Bourdel, N. et al., 2014) and incidence of early complications and side effects.

The secondary outcome will include the duration of sensory block, the time and the amount of post-procedure analgesic requirement, itching and any associated complications.

We hypothesized that CT guided ganglion impar block will be a good choice in pain reduction in patients with chronic pelvic pain. Pain reduction will be greater in dexamethasone and ketorolac group compared to alcohol group.Preinterventional assessment includes general, pain specific history taking (location, quality, intensity, relieving and provoking incidences) and pain in specific physical examination (inspection and palpation) will be carried out. Type of pelvic tumor, investigation related to tumor, previous operations, chemotherapy, basic demographic variables including age, sex and body mass index will be recorded. Routine investigations include bleeding profiles (bleeding time, clotting time, INR), blood picture, liver and kidney function tests will be carried out. A linear visual analogue scale (VAS) on a scale of 0-10 mm (where 0 for no pain and 10 for worst pain) will be explained to each patient. Written informed consent will be obtained, detailed information on risks and complications will be provided.The vital signs (heart rate, blood pressure, spo2) will be recorded. After establishing an access to peripheral venous line, 500 ml normal saline will be given to the patient, the patient will be in the prone position with a pillow under the abdomen to allow flexion of the lumbo-sacral spine with internal rotation of the lower extremities.All patients will be asked to empty the bladder and rectum before the start of the procedure to facilitate needle placement and avoid inadvertent injection. The pre-injection planning images will be obtained using CT with 2 mm axial section thickness. A needle localizer will be placed on the skin surface to identify and mark the sacro-coccygeal disc.

Sterilization of The patient's sacral and gluteal areas will be provided with povidone iodine antiseptic solution and this area was circumferentially draped with sterile towels. Under aseptic technique, a skin wheal will be raised with 2 ml lignocaine 0.5% using 23 G needle either in midline or paramedian approach. After identifying the ganglion impar, usually at the level of the sacro-coccygeal disc, a 25 G, 9 cm long spinal needle will be introduced at approximately 6-9 cm from midline and a small amount of non-ionic contrast medium (0.5 ml iopamidol; 300 mg/ml) will be injected. The midline approach may be selected according to patient position and operative condition. In the midline approach the sacro-coccygeal disc is identified and needle will be introduced perpendicular through the disc and just encroaching upon presacro-coccygeal space. The patient will be rescanned to confirm the position of the tip of the spinal needle at the anterior aspect of the sacro-coccygeal junction in the retroperitoneal space (Datir A and Connell D., 2010).

Thereafter, 3 ml lidocaine 2% will be injected, three minutes later 5 ml absolute alcohol 95% ± 8 mg dexamethasone or (15 mg ketorolac) will be slowly injected for therapeutic chemical neurolysis.

ELIGIBILITY:
Inclusion Criteria:

* patients of either sex aged between 20 to 70 years old with pelvic tumor

Exclusion Criteria:

* Patient's refusal.
* Sever Hepatic and renal impairment.
* History of allergy to the used drugs.
* Infection at the area of injection.
* Coagulopathies.

Ages: 20 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2018-07-01 (Actual); Primary Completion 2019-07-01 (Actual); Study Completion 2019-10-01 (Actual)

PRIMARY OUTCOMES:
the onset of sensory block | one week
  occurance of analgesia
patient satisfaction | 6 month
  patient satisfaction score ( Jones KD, Sutton C., 2003) by questionnaire for 100
intensity of pain | 6 month
  visual analogue scale (VAS) scale from 0 to 10 o no pain 10 maximum pain 0 better 10 worst
incidence of early complications | 6 month
  Early complications will be recorded including allergy, bleeding, hematoma, infection, perforation of the rectum and/or bowel, bladder incontinence and nerve root injury. The cauda equine syndrome is another potential complication

SECONDARY OUTCOMES:
the time and the amount of post-procedure analgesic requirement | 6 month
  the amount and timing of analgesic consumption and types of analgesics

CONTACTS AND LOCATIONS:
Overall Officials: Tarek M. Shams, MD, Study Director — : Professor of Anesthesia and Surgical Intensive Care
Locations (1):
- Mansoura university , oncology mansoura university center, Al Mansurah, Dakahlia Governorate, Egypt

IPD SHARING:
Plan to Share IPD: No